CLINICAL TRIAL: NCT04820972
Title: Early-Start Antiplatelet Treatment After Neurosurgery in Patients With Spontaneous Intracerebral Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: The Second Affiliated Hospital of Kunming Medical University (Other); First Affiliated Hospital of Fujian Medical University (Other); Second Xiangya Hospital of Central South University (Other); First Affiliated Hospital of Harbin Medical University (Other); Gangzhou Red Cross Hospital ，Jinan University (Unknown); Beijing Chao Yang Hospital (Other); RenJi Hospital (Other); Sichuan Academy of Medical Sciences (Other); Chongqing General Hospital (Other); Binzhou Medical University (Other); Fujian Medical University Union Hospital (Other); Shanxi Provincial People Hospital (Unknown); Beijing Friendship Hospital (Other); Qilu Hospital of Shandong University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Wang Shuo, Director of Department of Cerebrovascular Neurosurgery, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HX-A-007（2021）
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2023-06

CONDITIONS: Spontaneous Intracerebral Hemorrhage
Keywords: antiplatelet treatment; spontaneous intracerebral hemorrhage; early-start; neurosurgery
MeSH Terms: interventions — Platelet Aggregation Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- E-STAR group (Experimental)
  Interventions: Drug: Antiplatelet Agents
- traditional group (No Intervention)

INTERVENTIONS:
Drug: Antiplatelet Agents — using antiplatelet agents in 3 days after surgery
  Arms: E-STAR group

SUMMARY:
This study is a multicenter, prospective, open-label, endpoint-blind, randomized controlled study.Patients receiving surgical treatment for SICH were divided into groups using the random machine method. In addition to conventional treatment for spontaneous intracerebral hemorrhage, patients in the group of early initiation of antiplatelet therapy were given conventional dose of aspirin (100mg, qd) antiplatelet therapy starting from the 3rd day after surgery.An independent group of investigators evaluated cardiac, cerebral and peripheral vascular events and bleeding events at four different time points.To evaluate the benefits and safety of early postoperative initiation of antiplatelet therapy in patients with spontaneous intracerebral hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old.
* nontraumatic spontaneous intracerebral hemorrhage.
* postoperative patients with high risk of MACCPE:(1)previous history of cerebral infarction or TIA. (2)previous history of coronary heart disease or myocardial infarction.(3) use ASCVD Risk Estimator Plus（http://tools.acc.org/ASCVD-Risk-Estimator-Plus/#!/calculate/estimate/） to assess the risk of ischemic events for patients with no previous history of cerebral infarction, TIA, or coronary heart diseases or myocardial infarction,10 years risk>10% is defined as a high risk of cardiovascular ischemic events(4)The Caprini Risk Scale is used to assess the risk of venous thrombosis in the lower extremities.Score>2 is defined as a high risk of venous thrombosis.
* patients who received neurosurgical procedures to remove the hematoma, including craniotomy, endoscopic hematoma removal and hematoma aspiration.
* patients who signed informed consent.
* no history of allergy to salicylic acid preparation.
* patients who complete the preintervention assessment and meet the fellow criteria:(1)postoperative head CT showed no new infarction or hemorrhage(2)postoperative venous ultrasound of the lower extremity did not reveal deep vein thrombosis.(3)postoperative electrocardiogram and myocardial enzyme examination did not show acute myocardial ischemia or myocardial infarction.

Exclusion Criteria:

* there are structural cerebrovascular lesions (such as intracranial aneurysms, cerebrovascular malformations, etc.) or tumors in the area of bleeding or the bleeding is suspected to be related to these lesions.
* ischemic stroke with hemorrhagic conversion.
* secondary bleeding due to venous embolism.
* the malignant tumor is expected to have a survival of no more than 3 months.
* take antithrombotic agents((Vitamin K antagonists (warfarin) new anticoagulants(Dabigatun Rivaroxaban))) in addition to antiplatelet agents.
* previous history of thrombocytopenia or coagulation disorders.
* previous history of atrial fibrillation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
rate of intracranial hemorrhage | 7 days after surgery
rate of intracranial hemorrhage | 14 days after surgery
rate of intracranial hemorrhage | 30 days after surgery
rate of intracranial hemorrhage | 90 days after surgery
rate of major adverse cardiac/cerebrovascular and peripheral vessel events | 7 days after surgery
rate of major adverse cardiac/cerebrovascular and peripheral vessel events | 14 days after surgery
rate of major adverse cardiac/cerebrovascular and peripheral vessel events | 30 days after surgery
rate of major adverse cardiac/cerebrovascular and peripheral vessel events | 90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Wang, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Capital Medical University Affiliated Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Liu Q, Mo S, Wu J, Tong X, Wang K, Chen X, Chen S, Guo S, Li X, Li M, Peng L, Sun X, Wang Y, Sun J, Pu J, Zheng K, Zhang J, Liu Y, Yang Y, Wen Z, Nie X, Feng Y, Lan C, Tang H, Wang N, Li J, Miao Z, Lu X, Ning B, Zhao B, Kang D, Chen X, Zhang Y, Zhang Y, Wang A, Zhu C, Araki Y, Uda K, Yoshimura S, Uchida K, Morimoto T, Yoshioka H, Hasan D, Du R, Levitt MR, Cao Y, Wang S, Zhao J; E-start collaborators. Safety and efficacy of early versus delayed acetylsalicylic acid after surgery for spontaneous intracerebral haemorrhage in China (E-start): a prospective, multicentre, open-label, blinded-endpoint, randomised trial. Lancet Neurol. 2024 Dec;23(12):1195-1204. doi: 10.1016/S1474-4422(24)00424-1. PMID 39577920
- [Derived] Cochrane A, Chen C, Stephen J, Ronning OM, Anderson CS, Hankey GJ, Al-Shahi Salman R. Antithrombotic treatment after stroke due to intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Jan 26;1(1):CD012144. doi: 10.1002/14651858.CD012144.pub3. PMID 36700520
- [Derived] Wang K, Mo S, Liu Q, Pu J, Huang X, Kang D, Lin F, Zou D, Sun X, Ren J, Tong X, Li J, Salman RA, Wang N, Guo S, Liu Y, Zhang Y, Li X, Wu J, Wang S. Early-start antiplatelet therapy after operation in patients with spontaneous intracerebral hemorrhage and high risk of ischemic events (E-start): Protocol for a multi-centered, prospective, open-label, blinded endpoint randomized controlled trial. Front Aging Neurosci. 2022 Nov 23;14:1020224. doi: 10.3389/fnagi.2022.1020224. eCollection 2022. PMID 36506468